CLINICAL TRIAL: NCT06786897
Title: Expectations of Patients in Palliative Situation and Their Caregivers Concerning Blood Cell Transfusions in Haematology Department
Brief Title: Expectations of Patients in Palliative Situation
Acronym: ERAPH
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL24_0289; 2024-A02148-39 (Other: ANSM)
Record Dates: First submitted 2025-01-10; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: haematology; palliative situation
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient: Patient in palliative situation
  Interventions: Other: Questionnaire and Physical Exam

INTERVENTIONS:
Other: Questionnaire and Physical Exam — Questionnaires evaluating the expectations of patients in palliative situation, of paramedics and medical staff, concerning blood cell transfusions.

SUMMARY:
To date, there is a lack of data about the benefit of blood cell transfusions for patients diagnosed of a hematologic malignancy who are not eligible for curative treatments. Furthermore, there is no clear guideline about how to transfuse these patients and when the blood cell transfusions should be stopped.

Allogenic stem cell transplantation is nowadays the only curative treatment for patients with high-risk myeloid neoplasms. Knowing that the median age at diagnostic for acute myeloid leukemia is 68 years and this incidence increases after 65 years, a lot of patients won't be eligible for allogenic stem cell transplantation.

Besides, patients with haematologic malignancies are prone to cytopenias, due to their pathology and the treatments used to limit its progression. A study estimate that these patients need a median of 4 blood cell units per month, and it is known that repeated transfusions are associated with an increased risk of dying in hospital.

Finally, it is estimate that there was a lack of 20 000 blood cell units in France in 2022.

It therefore seems essential to find ways to optimize blood transfusion prescriptions in this population of patients who won't be eligible for curative treatments, with the main idea of maintaining or even improving their quality of life.

The investigators will study the expectations of patients in palliative situation, paramedics and medical staff concerning blood cell transfusions, by asking them if whether or not they believe that the transfusion planed to be administer will benefit the patient. To do this, investigators will distribute questionnaires before each blood cell transfusions to patients who will be included, to the paramedic who administered the transfusion and to the physician who prescribed the transfusion.

It is to investigators knowledge the first study to compare the expectations of patients in palliative situation, paramedics and medical staff concerning blood cell transfusions in hematology department, and follow the evolution of these expectations prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or more AND
* Diagnosed of an intermediate or high-risk acute leukemia and not eligible for allogenic stem cell transplantation Or
* Diagnosed of a high-risk myelodisplasic syndrome and not eligible for allogenic stem cell transplantation Or
* Diagnosed of an intermediate or high-risk myelofibrosis and not eligible for allogenic stem cell transplantation Or
* Diagnosed of a chronic myeloid leukemia in blast crisis phase and not eligible for allogenic stem cell transplantation Or
* Relapsing after allogenic stem cell transplantation and not eligible for a second allogenic stem cell transplantation

Exclusion criteria:

* Patients who can't read
* Patients who can't write
* Patients who can't express their consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruted in palliative department of the hospital
Sampling Method: Non-Probability Sample
Enrollment: 37 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the benefit of blood cell transfusion before each blood cell transfusion | up to 52 weeks
  Evaluate the concordance for the perceptions of the benefit of blood cell transfusions in a palliative situation in hematology department between patients, paramedical and medical staff

SECONDARY OUTCOMES:
Number of days before death | through study completion, an average of 1 year
  Define the median number of days before death, from which patients believe they no longer benefit from blood transfusions

CONTACTS AND LOCATIONS:
Locations (1):
- UH Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Yes
Publication of the results
Supporting Information: CSR
Access Criteria: Publication